CLINICAL TRIAL: NCT02528526
Title: A Phase IB/IIA, Single-centered Study of the Effects of OXY111A in Primary and Secondary Hepato-Pancreato-Biliary Neoplasia
Brief Title: Effects of OXY111A in Primary and Secondary Hepato-Pancreato-Biliary Neoplasm
Acronym: OXY1A
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXY1A_2014-0374
Record Dates: First submitted 2014-11-11; First posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Pancreatic Neoplasms; Hepatocellular Cancer; Cholangiocarcinoma; Colorectal Neoplasms
Keywords: Hypoxia; Pancreatic Neoplasms; Hepatocellular Cancer; Cholangiocarcinoma; Colorectal Neoplasms; Treatment
MeSH Terms: conditions — Pancreatic Neoplasms; Liver Neoplasms; Cholangiocarcinoma; Colorectal Neoplasms; Hypoxia | interventions — inositol trispyrophosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Add-on application of Myo-inositol trispyrophosphate, total of 9 times, 3 applications per week, over 3 weeks.
  Interventions: Drug: OXY111A

INTERVENTIONS:
Drug: OXY111A — OXY111A intravenous infusion
  Other Names: Myo-inositol trispyrophosphate

SUMMARY:
The purpose of the study is to evaluate whether the novel anti-cancer drug OXY111A is safe and tolerated in patients with primary and secondary hepato-pancreato-biliary and gastrointestinal neoplasia as measured by exploring the maximum tolerated dose (MTD). At level of MTD, additional patients will be included aimed for assessing the efficacy profile in these neoplasia entities.

DETAILED DESCRIPTION:
The IMP OXY111A counteracts hypoxia-induced tumor aggressiveness showing decreased tumor burden and increased survival in five different animal solid tumor models both applied as monotherapy and increased beneficial effects when followed by standard chemotherapy. The unique ability of the IMP counteract hypoxic tumor behaviour along with its non-toxic side effects tested both in animals and healthy volunteers is of outmost interest to explore in patients with solid tumors.

The study seeks primarily to determine the safety and tolerability of OXY111A in patients with primary and secondary hepato-pancreato-biliary and gastrointestinal neoplasia as measured by exploring the MTD in a conservative 3+3 dose escalation schedule. The window for DLT assessment is from first dose of study drug until first dose of standard of care chemotherapy or 10 days following completion of last dose of study drug (whichever is shorter in duration). Additionally, we will assess efficacy of OXY111A on decreasing tumor volume, metabolic activity, as well as circulatory tumor and angiogenic markers.

ELIGIBILITY:
Inclusion Criteria:

* Study Indication: patients diagnosed for non-resectable hepato-pancreato-biliary or gastrointestinal neoplasm
* Male and Female patients ≥ 18 years of age
* Signed Informed Consent after being informed
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≥ 2 at study entry.
* A life-expectancy of >3 months
* Adequate hematologic and renal function
* Use of effective contraception (per the institutional standard), if procreative potential exists
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 28 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy (palliative radiation therapy is allowed)
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by collection of adverse effects information | 10 weeks
  Safety variables and patient tolerance as measured by collection of adverse effects information according to Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
Efficacy as measured by FDG-PET scan | 5 months
  Assessment of tumor response with 18F-FDG PET in FDG-avid tumors using EORTC criteria
Efficacy as measured by MRI | 5 months
  Assessment of tumor response with MRI in non-FDG-avid tumors using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain, Clavien, Principal Investigator — University Hospital Zurich, Visceral Surgery
Locations (1):
- University Hospital Zurich, Visceral Surgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Aprahamian M, Bour G, Akladios CY, Fylaktakidou K, Greferath R, Soler L, Marescaux J, Egly JM, Lehn JM, Nicolau C. Myo-InositolTrisPyroPhosphate treatment leads to HIF-1alpha suppression and eradication of early hepatoma tumors in rats. Chembiochem. 2011 Mar 21;12(5):777-83. doi: 10.1002/cbic.201000619. Epub 2011 Mar 2. PMID 21370375
- [Background] Derbal-Wolfrom L, Pencreach E, Saandi T, Aprahamian M, Martin E, Greferath R, Tufa E, Choquet P, Lehn JM, Nicolau C, Duluc I, Freund JN. Increasing the oxygen load by treatment with myo-inositol trispyrophosphate reduces growth of colon cancer and modulates the intestine homeobox gene Cdx2. Oncogene. 2013 Sep 5;32(36):4313-8. doi: 10.1038/onc.2012.445. Epub 2012 Oct 8. PMID 23045284
- [Background] Kieda C, El Hafny-Rahbi B, Collet G, Lamerant-Fayel N, Grillon C, Guichard A, Dulak J, Jozkowicz A, Kotlinowski J, Fylaktakidou KC, Vidal A, Auzeloux P, Miot-Noirault E, Beloeil JC, Lehn JM, Nicolau C. Stable tumor vessel normalization with pO(2) increase and endothelial PTEN activation by inositol trispyrophosphate brings novel tumor treatment. J Mol Med (Berl). 2013 Jul;91(7):883-99. doi: 10.1007/s00109-013-0992-6. Epub 2013 Mar 9. PMID 23471434
- [Background] Raykov Z, Grekova SP, Bour G, Lehn JM, Giese NA, Nicolau C, Aprahamian M. Myo-inositol trispyrophosphate-mediated hypoxia reversion controls pancreatic cancer in rodents and enhances gemcitabine efficacy. Int J Cancer. 2014 Jun 1;134(11):2572-82. doi: 10.1002/ijc.28597. Epub 2013 Nov 25. PMID 24214898
- [Background] Fylaktakidou KC, Lehn JM, Greferath R, Nicolau C. Inositol tripyrophosphate: a new membrane permeant allosteric effector of haemoglobin. Bioorg Med Chem Lett. 2005 Mar 15;15(6):1605-8. doi: 10.1016/j.bmcl.2005.01.064. PMID 15745806
- [Derived] Schneider MA, Linecker M, Fritsch R, Muehlematter UJ, Stocker D, Pestalozzi B, Samaras P, Jetter A, Kron P, Petrowsky H, Nicolau C, Lehn JM, Humar B, Graf R, Clavien PA, Limani P. Phase Ib dose-escalation study of the hypoxia-modifier Myo-inositol trispyrophosphate in patients with hepatopancreatobiliary tumors. Nat Commun. 2021 Jun 21;12(1):3807. doi: 10.1038/s41467-021-24069-w. PMID 34155211
- [Derived] Limani P, Linecker M, Kron P, Samaras P, Pestalozzi B, Stupp R, Jetter A, Dutkowski P, Mullhaupt B, Schlegel A, Nicolau C, Lehn JM, Petrowsky H, Humar B, Graf R, Clavien PA. Development of OXY111A, a novel hypoxia-modifier as a potential antitumor agent in patients with hepato-pancreato-biliary neoplasms - Protocol of a first Ib/IIa clinical trial. BMC Cancer. 2016 Oct 19;16(1):812. doi: 10.1186/s12885-016-2855-3. PMID 27756258
- See also: Swiss Hepato-Pancreato-Biliary (HPB) Center, University Hospital Zurich, Switzerland — http://www.hpb-center.ch